CLINICAL TRIAL: NCT02878252
Title: A Cross-sectional Study to Determine the Proportion and Clinical Characteristics of COPD Patients With Asthma Symptoms in Asia (ACOS) and Describe Current Practices in Diagnosis and Management
Brief Title: Non-interventional Study of COPD Patients With Asthma Overlap Syndrome in Viet Nam and Taiwan
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ASK CRE Private Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: D2287R00106
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Patients With Asthma-COPD Overlap Syndrome (ACOS)
Keywords: COPD, Asthma, ACOS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study to determine the proportion and clinical characteristics of COPD patients with asthma symptoms (ACOS) and describe current practices in diagnosis and management in Viet Nam and Taiwan.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of chronic morbidity and mortality. Around 15% to 20% of COPD patients would present with features of asthma and are considered to have the overlap syndrome of COPD and asthma, commonly called asthma-COPD overlap syndrome (ACOS). In Asia, specifically Taiwan, the overall prevalence of ACOS in patients with COPD is approximately 17.4%. COPD patients with asthma symptoms represent a relevant clinical population because they have worse health-related quality of life.

Given the increased morbidity among COPD patients with asthma overlap, it is critical that these patients are properly characterized to aid the appropriate diagnosis and treatment. The Global Initiative for Asthma (GINA) and Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines have given joint recommendations on the identification, diagnosis and treatment of these patients. These recommendations have been adapted for use in the Asia Area countries. The primary objective of this study is to determine the proportion and clinical characteristics of patients with ACOS as defined by the joint GINA and GOLD recommendation amongst diagnosed COPD patients seen at the out-patient clinics.

This study is planned to determine the proportion of patients with ACOS as defined by the joint GINA and GOLD recommendation amongst diagnosed COPD patients seen at the out-patient clinics

ELIGIBILITY:
Inclusion Criteria:

* All patients with confirmed diagnosis of COPD {post-bronchodilator FEV1/FVC<0.7 (FEV1 - forced expiratory volume at one second, FVC - forced vital capacity) based on the medical records}
* Aged >40 years old at time of diagnosis
* Seen at out-patient clinic

Exclusion Criteria:

* Patients currently with acute exacerbation of COPD by GOLD definition (any worsening of a patient's respiratory symptoms that is beyond normal day-to-day variations and requires a change in medication)
* Patients with respiratory diseases that can show similar symptoms to chronic airway diseases such as bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, endobronchial TB, and lung cancer, or those who have history of these diseases based on physician's judgment
* Patients currently diagnosed with pneumonia and acute bronchitis
* Patients currently randomized in other clinical studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with COPD who are seen at the outpatient clinics of Pulmonary Specialists
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
proportion of ACOS patients among COPD-diagnosed patients seen at the out-patient clinics | 6 month
  To determine the proportion and clinical characteristics of patients with Asthma-COPD Overlap Syndrome (ACOS) as defined by the joint GINA and GOLD recommendation amongst diagnosed COPD patients seen at the out-patient clinic.

SECONDARY OUTCOMES:
symptom control assessment | 6 months
  To review the current practices of symptom control assessment

OTHER OUTCOMES:
medications given to ACOS patients in current practice | 6 months
  To review the medications given to COPD patients with asthma compared to guideline recommendations

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (3):
  - Research Site, Kaohsing
  - Research Site, Taichung
  - Research Site, Taipei
- Vietnam (2):
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3988&filename=CSR_synopsis_(ACOS_NIS_Study)TWVN.pdf